CLINICAL TRIAL: NCT02825290
Title: Modified Luteal Support for Frozen-Thawed Embryo Transfer - A Prospective Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Eran Zilberberg, Doctor, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2537-15-SMC
Record Dates: First submitted 2016-07-03; First posted 2016-07-07 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Embryo Transfer; Luteal Support
Keywords: Frozen-thawed embryo transfer (FET); Luteal support; Progesterone; Natural cycle; Cryopreservation; IVF; hCG; GnRH-Agonist; Pregnancy rate
MeSH Terms: interventions — Chorionic Gonadotropin; Ovidrel; Triptorelin Pamoate; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): hCG (Choriogonadotropin alfa; Ovitrelle 250 mcg) on day of embryo transfer & GnRH-agonist (Triptorelin acetate; Decapeptyl 0.1 mg) after 4 days In addition to the usual progesterone luteal support.
  Interventions: Drug: Choriogonadotropin alfa; Drug: Triptorelin acetate
- Control group (No Intervention): The usual progesterone only luteal phase support.

INTERVENTIONS:
Drug: Choriogonadotropin alfa
  Other Names: recombinant hCG; Ovitrelle; Ovidrel
  Arms: Study group
Drug: Triptorelin acetate
  Other Names: GnRH-Agonist; Decapeptyl
  Arms: Study group

SUMMARY:
This study evaluates the outcomes of frozen-thawed embryo transfer (FET) success rate with modified luteal support - addition of a single injection of HCG and GnRH-agonist, on day of ET and 4 days later, respectively vs. traditional luteal support with vaginal progesterone only in ovulating women.

DETAILED DESCRIPTION:
Background With the recent trend toward single embryo transfer (ET) adopted in an attempt to reduce the risk of multiple pregnancy, the remaining extra embryos are cryopreserved, providing further possibilities for conception after the initial fresh transfer. Moreover, several studies that compared fresh and frozen-thawed embryo transfer (FET) cycles in normal responders have demonstrated a significantly higher clinical pregnancy rate per transfer in the FET versus the fresh cycles.

There are several currently employed replacement protocols for FET. The choice of protocol depends on the individual woman's ovarian function and convenience of the method, as well as on the experience gained with the method by the physicians. Whatever protocol is used, the success requires optimal synchronization between the embryonic stage at thawing and date of the endometrium within the endometrial preparation cycle. While there is a consensus regarding the duration, route of delivery and dosage of estrogen supplementation, and the optimal ultrasonographic endometrial appearance and thickness, the effect of the different modes of luteal support remains unclear.

Prompted by the study demonstrating higher ongoing pregnancy rate following the transfer of frozen-thawed embryos in natural cycles with spontaneous LH rise compared with natural cycles controlled by hCG for final oocyte maturation and the reports showing improved pregnancy rate in patients who received a mid-luteal injection of a GnRH-agonist (0.1 mg triptorelin), the investigators started beginning at June 2014 to offer ovulatory patients with regular menstrual cycles a natural FET with modified luteal support. Starting on the day of spontaneous ovulation, patients received daily vaginal progesterone, supplemented by a single injection of HCG and GnRH-agonist, on day of ET and 4 days later, respectively.

The results for this study were very promising - the investigators were able to show a significant increase in implantation rate (30% vs. 17%; p<0.03), clinical pregnancy (48% vs. 26%; p<0.01) and ongoing pregnancy (39% vs. 20%; p<0.01) for the patients receiving the aforementioned modified luteal support protocol.

After the completion of this retrospective study the investigators are heading to prove the superiority of the modified luteal support protocol for ovulatory patients by conducting a prospective study.

Materials & Methods Study design - A prospective, randomized, blinded study. Primary endpoint - Ongoing pregnancy. Secondary endpoints - Implantation rate, clinical pregnancy. Study sample - According to the previous, retrospective study the investigators will need 31 patients in each study arm in order to show an increase from 20% clinical pregnancy to 39% (confidence level 5%, beta error level 50%).

The patients - The investigators will offer each patient treated in the unit for frozen-thawed embryo transfer to participate in the study. The randomization of the participants will be on the day of embryo transfer with a computer program on a 1:1 enrollment ratio.

All transfers will be performed by an experienced physician who will be blinded to the luteal support protocol.

Both groups will be treated with the accepted progesterone luteal support - starting on ovulation day - vaginal progesterone 90 mg (Crinone; Merck Serono, Hellerup, Denmark) once a day.

Study group - Patients in the study group will receive additional two injections - the first - recombinant hCG 250 mcg (Ovitrelle; Merck Serono) on the transfer day and the second - GnRH-agonist 0.1 mg (Decapeptyl; Ferring Pharmaceuticals Israel) 4 days after the embryo transfer day. Patients in the control group will receive no injection.

B-hCG levels will be examined 12 days after embryo transfer and if positive ultrasound examinations will be performed as usual to document pregnancy outcome.

The data - The investigators will use demographic data such as age, BMI, gynecological data as gravida, para, etiology of infertility and data about previous & current IVF treatments such as number of treatments, stimulation protocol, hormone levels, number of oocytes, embryos' characteristics, etc.

Statistics - Statistical analysis will be performed with Student's t-test and Chi square, as appropriate. Results will be presented as means ± standard deviations; p<0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years old women
* Spontaneously ovulating women
* Treated in our IVF unit for frozen-thawed embryo transfer
* At least one top quality embryo

Exclusion Criteria:

* PGD patients
* More than 4 previous embryo transfers

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy | About 10-12 weeks after embryo transfer
  Number of viable pregnancies at about 10-12 weeks of gestation.

SECONDARY OUTCOMES:
Implantation rate | 2 weeks after embryo transfer
  Positive BhCG blood test
Clinical pregnancy | About 3-4 weeks after embryo transfer
  Visible intrauterine gestational sacs on ultrasound exam

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thurin A, Hausken J, Hillensjo T, Jablonowska B, Pinborg A, Strandell A, Bergh C. Elective single-embryo transfer versus double-embryo transfer in in vitro fertilization. N Engl J Med. 2004 Dec 2;351(23):2392-402. doi: 10.1056/NEJMoa041032. PMID 15575055
- [Background] Le Lannou D, Griveau JF, Laurent MC, Gueho A, Veron E, Morcel K. Contribution of embryo cryopreservation to elective single embryo transfer in IVF-ICSI. Reprod Biomed Online. 2006 Sep;13(3):368-75. doi: 10.1016/s1472-6483(10)61441-1. PMID 16984767
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C. Clinical rationale for cryopreservation of entire embryo cohorts in lieu of fresh transfer. Fertil Steril. 2014 Jul;102(1):3-9. doi: 10.1016/j.fertnstert.2014.04.018. Epub 2014 May 17. PMID 24842675
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C, Thomas S. Evidence of impaired endometrial receptivity after ovarian stimulation for in vitro fertilization: a prospective randomized trial comparing fresh and frozen-thawed embryo transfer in normal responders. Fertil Steril. 2011 Aug;96(2):344-8. doi: 10.1016/j.fertnstert.2011.05.050. Epub 2011 Jul 6. PMID 21737072
- [Background] Orvieto R, Fisch B, Feldberg D. Endometrial Preparation for Patients undergoing Frozen- Thawed Embryo Transfer Cycles. In: The Art & Science of Assisted Reproductive Techniques. G. Allahbadia, R. asuray, R. Merchant, Eds. Jaypee Brothers Medical Publishers (P) Ltd. New Delhi, India, 2003, pp. 396-9.
- [Background] Navot D, Laufer N, Kopolovic J, Rabinowitz R, Birkenfeld A, Lewin A, Granat M, Margalioth EJ, Schenker JG. Artificially induced endometrial cycles and establishment of pregnancies in the absence of ovaries. N Engl J Med. 1986 Mar 27;314(13):806-11. doi: 10.1056/NEJM198603273141302. PMID 3951513
- [Background] Pritts EA, Atwood AK. Luteal phase support in infertility treatment: a meta-analysis of the randomized trials. Hum Reprod. 2002 Sep;17(9):2287-99. doi: 10.1093/humrep/17.9.2287. PMID 12202415
- [Background] Meldrum DR. Female reproductive aging--ovarian and uterine factors. Fertil Steril. 1993 Jan;59(1):1-5. doi: 10.1016/s0015-0282(16)55608-8. PMID 8419194
- [Background] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333
- [Background] Tesarik J, Hazout A, Mendoza C. Enhancement of embryo developmental potential by a single administration of GnRH agonist at the time of implantation. Hum Reprod. 2004 May;19(5):1176-80. doi: 10.1093/humrep/deh235. Epub 2004 Apr 7. PMID 15070873
- [Background] Tesarik J, Hazout A, Mendoza-Tesarik R, Mendoza N, Mendoza C. Beneficial effect of luteal-phase GnRH agonist administration on embryo implantation after ICSI in both GnRH agonist- and antagonist-treated ovarian stimulation cycles. Hum Reprod. 2006 Oct;21(10):2572-9. doi: 10.1093/humrep/del173. Epub 2006 Aug 22. PMID 16926261
- [Background] Orvieto R, Brengauz M, Feldman B. A novel approach to normal responder patient with repeated implantation failures--a case report. Gynecol Endocrinol. 2015 Jun;31(6):435-7. doi: 10.3109/09513590.2015.1005595. Epub 2015 Mar 3. PMID 25731193
- [Background] Haas J, Lantsberg D, Feldman N, Manela D, Machtinger R, Dar S, Rabinovici J, Orvieto R. Modifying the luteal phase support in natural cycle frozen-thawed embryo transfer improves cycle outcome. Gynecol Endocrinol. 2015;31(11):891-3. doi: 10.3109/09513590.2015.1075502. Epub 2015 Aug 18. PMID 26288149